CLINICAL TRIAL: NCT00961974
Title: Intensive Care Program for Youth With Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Charles H. Hood Foundation (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lori Laffel, Chief, Pediatric, Adolescent, & Young Adult Section; Investigator, Genetics & Epidemiology Section, Joslin Diabetes Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-06; R01DK046887 (NIH)
Record Dates: First submitted 2009-08-18; First posted 2009-08-19 (Estimated); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Type 1 Diabetes
Keywords: type 1 diabetes; hemoglobin A1c; family; involvement; responsibility; conflict; quality of life; children
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Margins of Excision

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard Care (No Intervention): * Routine diabetes support and education from diabetes health care team
  * Assistance from a non-medical case manager (Care Ambassador) to schedule appointments, provide reminders about appointments, and help families contact health care providers about questions or concerns
- Care Plus (Experimental): * Routine diabetes support and education from diabetes health care team
  * Assistance from a non-medical case manager (Care Ambassador) to schedule appointments, provide reminders about appointments, and help families contact health care providers about questions or concerns
  Interventions: Behavioral: Care Ambassador Intervention
- Care Ultra (Experimental): * Routine diabetes support and education from diabetes health care team
  * Assistance from a non-medical case manager (Care Ambassador) to schedule appointments, provide reminders about appointments, and help families contact health care providers about questions or concerns
  Interventions: Behavioral: Care Ambassador Intervention; Behavioral: Psychoeducational Intervention

INTERVENTIONS:
Behavioral: Care Ambassador Intervention — Care Ambassador provides additional monthly outreach (by phone or e-mail) to families between clinic visits.
  Arms: Care Plus; Care Ultra
Behavioral: Psychoeducational Intervention — A psychoeducational intervention module is reviewed with the family by the Care Ambassador at each clinic visit. The intervention focuses on incorporating intensive therapy into the daily routine of the child through positive family support for blood glucose monitoring and healthy eating. The intervention modules review positive family communication, realistic expectations, ways to avoid perfectionism and maintain family involvement, prevention of hypoglycemia, avoidance of diabetes-specific family conflict, and approaches to reducing "diabetes burnout".
  Arms: Care Ultra

SUMMARY:
The purpose of this study was to determine the ability of a family-focused, office-based intervention to improve medical and behavioral outcomes for children and adolescents with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Age 8-16 years
* Type 1 diabetes diagnosed by standard American Diabetes Association criteria
* Type 1 diabetes duration of at least 6 months
* Residence in northeastern U.S.
* Established clinic patient
* Fluency in English or Spanish

Exclusion Criteria:

* Major psychiatric disorder (e.g., major depression, severe eating disorder, mental retardation)
* Unstable living environment (e.g., Department of Social Services or Department of Youth Services involvement)

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2002-04; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Glycemic control, assessed by hemoglobin A1c | Every 3 months

SECONDARY OUTCOMES:
Psychosocial factors (diabetes-specific family conflict, responsibility-sharing for diabetes management tasks, quality of life, affect regarding blood glucose monitoring, disordered eating behaviors) | Annually
Weight, assessed by z-BMI (age- and gender-adjusted body mass index) | Every 3 months
Frequency of hospitalizations, emergency department visits, and episodes of severe hypoglycemia | Every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lori Laffel, MD, MPH, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Butler DA, Zuehlke JB, Tovar A, Volkening LK, Anderson BJ, Laffel LM. The impact of modifiable family factors on glycemic control among youth with type 1 diabetes. Pediatr Diabetes. 2008 Aug;9(4 Pt 2):373-81. doi: 10.1111/j.1399-5448.2008.00370.x. PMID 18774997
- [Background] Svoren BM, Volkening LK, Butler DA, Moreland EC, Anderson BJ, Laffel LM. Temporal trends in the treatment of pediatric type 1 diabetes and impact on acute outcomes. J Pediatr. 2007 Mar;150(3):279-85. doi: 10.1016/j.jpeds.2006.12.009. PMID 17307546
- [Background] Moreland EC, Tovar A, Zuehlke JB, Butler DA, Milaszewski K, Laffel LM. The impact of physiological, therapeutic and psychosocial variables on glycemic control in youth with type 1 diabetes mellitus. J Pediatr Endocrinol Metab. 2004 Nov;17(11):1533-44. doi: 10.1515/jpem.2004.17.11.1533. PMID 15570991
- [Result] Katz ML, Volkening LK, Butler DA, Anderson BJ, Laffel LM. Family-based psychoeducation and Care Ambassador intervention to improve glycemic control in youth with type 1 diabetes: a randomized trial. Pediatr Diabetes. 2014 Mar;15(2):142-50. doi: 10.1111/pedi.12065. Epub 2013 Aug 5. PMID 23914987